CLINICAL TRIAL: NCT03739619
Title: A Phase I/II Study of Gemcitabine, Bendamustine, and Nivolumab in Patients With Relapsed or Refractory Classical Hodgkin Lymphoma
Brief Title: Gemcitabine, Bendamustine, and Nivolumab in Patients With Relapsed or Refractory Classical Hodgkin Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Bristol-Myers Squibb (Industry); National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Jonathon Cohen, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00104033; NCI-2018-02221 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Winship4388-18 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2018-11-01; First posted 2018-11-14 (Actual); Results first posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Recurrent Hodgkin Lymphoma; Refractory Hodgkin Lymphoma; Classical Hodgkin Lymphoma; Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — Bendamustine Hydrochloride; Gemcitabine; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Gemcitabine, bendamustine, nivolumab (Experimental): Patients receive gemcitabine IV over 30 minutes on day 1, bendamustine IV over 30 minutes on days 1 and 2, and nivolumab over 60 minutes IV on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients may then receive nivolumab IV over 60 minutes on day 1. Treatment with single agent nivolumab repeats every 28 days for up to 26 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bendamustine; Drug: Gemcitabine; Biological: Nivolumab

INTERVENTIONS:
Drug: Bendamustine — Given IV
  Other Names: Bendamustine Hydrochloride; Cytostasan Hydrochloride; Levact; Ribomustin; SyB L-0501; Treanda
Drug: Gemcitabine — Given IV
  Other Names: dFdC; dFdCyd; Difluorodeoxycytidine
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo

SUMMARY:
This phase I/II trial studies the side effects and best dose of gemcitabine, bendamustine, and nivolumab when given together and to see how well they work in treating patients with classic Hodgkin lymphoma that has come back or does not respond to treatment. Drugs used in chemotherapy, such as gemcitabine and bendamustine, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Immunotherapy with monoclonal antibodies, such as nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving gemcitabine, bendamustine, and nivolumab may work better in treating patients with classic Hodgkin lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the toxicity and determine the maximum tolerated dose (MTD) of combined gemcitabine, bendamustine, and nivolumab in patients with relapsed/refractory classical Hodgkin lymphoma.

II. To determine the efficacy of bendamustine, gemcitabine, and nivolumab in patients with relapsed/refractory classical Hodgkin lymphoma.

SECONDARY OBJECTIVES:

I. To evaluate the duration of response, progression-free survival, and overall survival for patients with relapsed/refractory classical Hodgkin lymphoma who receive gemcitabine, bendamustine, and nivolumab, including those who receive nivolumab maintenance.

OUTLINE: This is a phase I, dose-escalation study followed by a phase II study.

Patients receive gemcitabine intravenously (IV) over 30 minutes on day 1, bendamustine IV over 30 minutes on days 1 and 2, and nivolumab over 60 minutes IV on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients may then receive nivolumab IV over 60 minutes on day 1. Treatment with single agent nivolumab repeats every 28 days for up to 26 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented classical Hodgkin lymphoma that is recurrent or refractory after standard chemotherapy. Core biopsies are acceptable if they contain adequate tissue for primary diagnosis and immunophenotyping. Bone marrow biopsies as the sole means of diagnosis are not acceptable. At least one biopsy-proven relapse is required for enrollment, but patients who have multiply relapsed disease do not require repeat biopsy if not clinically indicated
* Prior treatment: patients must have relapsed or progressed after at least one prior therapy

  * Patients with relapsed or refractory disease following autologous stem cell transplantation are permitted. Due to the risk of treatment-refractory graft versus host disease (GVHD), patients who have previously completed an allogeneic transplant are excluded.
  * Patients may have received gemcitabine, bendamustine, or nivolumab in the past but may not have discontinued therapy due to toxicity felt to be related to that specific drug
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Measurable disease must be present either on physical examination or imaging studies. Non-measurable disease alone is not acceptable

  * Measurable disease

    * Lesions that can be accurately measured in at least two dimensions as ≥ 1.0 x 1.0 cm by computerized tomography (CT), positron emission tomography (PET)/CT (positron emission tomography/CT), or magnetic resonance imaging (MRI).
    * If identified by PET/CT, there must be at least one lesion that demonstrates abnormal fludeoxyglucose (FDG) avidity, consistent with active disease. Ultrasound or physical examination alone may not be utilized to confirm measurable disease
  * Non-measurable disease

    * All other lesions, including small lesions (less than 1.0 x 1.0 cm) and truly non-measurable lesions
    * Lesions that are considered non-measurable include the following:

      * Bone lesions (lesions if present should be noted)
      * Ascites
      * Pleural/pericardial effusion
      * Lymphangitis cutis/pulmonis
      * Bone marrow (involvement by Hodgkin lymphoma should be noted)
* Non-pregnant and non-nursing. Women and men of reproductive potential should agree to use an effective means of birth control
* Patients with human immunodeficiency virus (HIV) infection are eligible. Patients with HIV infection must meet the following: no evidence of co-infection with hepatitis B or C; cluster of differentiation 4+ (CD4+) count ≥ 400/mm; no evidence of resistant strains of HIV; on anti-HIV therapy with an HIV viral load < 50 copies HIV ribonucleic acid (RNA)/mL. Patients with HIV must have ongoing follow-up with an infectious disease specialist and must have been evaluated within 90 days of cycle 1 day 1
* Patients with a history of hepatitis C are eligible as long as the hepatitis C has been treated and cleared and they have no evidence of hepatic dysfunction related to hepatitis C. Patients must have been seen by a hepatologist within 6 months of cycle 1 day 1
* Patients who test positive for hepatitis B core antibody may enroll on the study as long as they test negative for both hepatitis B surface antigen and hepatitis B deoxyribonucleic acid (DNA), and if they have no evidence of hepatic dysfunction that is felt to be related to hepatitis B
* Patients must have adequate pulmonary function, defined as the following:

  * No history of drug-related, radiation-induced, or autoimmune pneumonitis requiring hospital admission
  * Baseline pulse oximetry reading of ≥ 92% on room air
  * Patients with a history of asthma or chronic obstructive pulmonary disease (COPD) must have no oxygen requirement, must have not had a hospital admission for COPD/asthma exacerbation within the past 2 years, and must not have received systemic steroids (≥ 10 mg prednisone for more than 7 days) for asthma/COPD within the past 2 years
* Patients with hypothyroidism or type 1 diabetes mellitus that are on chronic hormonal therapy and which are well-controlled are eligible
* Granulocytes ≥ 1000/µl
* Platelet count ≥ 75,000/µl
* Creatinine clearance ≥ 50 mL/min
* Bilirubin ≤ 2.0 mg/dL
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤ 2.0 x upper limits of normal

Exclusion Criteria:

* Due to the teratogenic potential of these agents, pregnant or nursing patients may not be enrolled
* Patients may not have an auto-immune disease requiring systemic immunosuppression, biologic therapy, and/or steroid use (≥ 10 mg daily of prednisone or equivalent)
* Patients with current or prior central nervous system (CNS) involvement with lymphoma are not eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2023-12-22 (Actual); Study Completion 2025-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathon Cohen, MD, MS, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gemcitabine, Bendamustine, Nivolumab
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Gemcitabine, Bendamustine, Nivolumab
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerable Dose (Phase I)
Description: Maximum tolerable dose will be defined as the highest dose level where at most 1 of 6 patients experience dose limiting toxicity (DLT).
Time Frame: Up to completion of course 2 at 42 days after study start
Population: The median values were not reached. No MTD events were observed within the trial time frame; thus, median MTD were not reached.
Measure: Count of Participants; unit: Participants
Arm/Group | Gemcitabine, Bendamustine, Nivolumab
Number analyzed (Participants) | 3
Participants | NA — The median values were not reached. No MTD events were observed within the trial time frame; thus, median MTD were not reached.

2. Primary Outcome: Complete Response (CR) Rate (Phase II)
Description: Complete response rate will be determined by dividing the number of CRs (per Lugano criteria) by the total number of evaluable patients.
Time Frame: Up to 2 years from discontinuation of study therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Gemcitabine, Bendamustine, Nivolumab
Number analyzed (Participants) | 2
Participants | 1

3. Secondary Outcome: Overall Response Rate (Phase II)
Description: Overall response rate will be evaluated using Lugano criteria of response. Overall response rate will be defined as the total number of patients achieving a partial response or CR as best response through cycle 6 divided by total number of patients treated.
Time Frame: Up to 2 years from discontinuation of study therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Gemcitabine, Bendamustine, Nivolumab
Number analyzed (Participants) | 2
Participants | 1

4. Secondary Outcome: Duration of Response (Phase II)
Description: Duration of response will be evaluated using Lugano criteria of response and will be determined from date of best response to progression or death.
Time Frame: Up to 2 years from discontinuation of study therapy
Measure: Mean (95% Confidence Interval); unit: Days
Arm/Group | Gemcitabine, Bendamustine, Nivolumab
Number analyzed (Participants) | 1
Days | 892

5. Secondary Outcome: Progression Free Survival (PFS) (Phase II)
Description: Progression free survival will be evaluated using Lugano criteria and will be determined from date of first dose of study drug to progression or death.
Time Frame: Up to 2 years from discontinuation of study therapy
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gemcitabine, Bendamustine, Nivolumab
Number analyzed (Participants) | 3
months | NA [NA to NA] — Too few events for a median to be reached. @ Timepoint 1.0 (NA,NA - not computable as no patient received an event) The median values were not reached. No PFS events were observed within the trial time frame; thus, median PFS were not reached.

6. Secondary Outcome: Overall Survival (OS) (Phase II)
Description: Overall survival will be evaluated using Lugano criteria and will be determined from date of first dose of study drug to death from any cause.
Time Frame: Up to 2 years from discontinuation of study therapy
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gemcitabine, Bendamustine, Nivolumab
Number analyzed (Participants) | 3
months | NA [NA to NA] — The median values were not reached. No OS events were observed within the trial time frame; thus, median OS were not reached.

ADVERSE EVENTS:
Time Frame: Adverse Events monitored/assessed up to 2 years. All-Cause Mortality monitored/assessed up to 2 years from discontinuation of study therapy a maximum of 4 years
Arm/Group | Gemcitabine, Bendamustine, Nivolumab
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 2/3
Other Adverse Events (participants affected / at risk) | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine, Bendamustine, Nivolumab (N=3)
Hospitalization (Respiratory, thoracic and mediastinal disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine, Bendamustine, Nivolumab (N=3)
Anemia (Blood and lymphatic system disorders) | 1 (5)
Decreased Platelet Count (Investigations) | 1 (3)
Headache (Nervous system disorders) | 2 (3)
Hypertension (Vascular disorders) | 1 (7)
Hypokalemia (Metabolism and nutrition disorders) | 1 (3)
Vomiting (Gastrointestinal disorders) | 1 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-07-05): https://cdn.clinicaltrials.gov/large-docs/19/NCT03739619/Prot_SAP_001.pdf
  • Informed Consent Form (2021-09-01): https://cdn.clinicaltrials.gov/large-docs/19/NCT03739619/ICF_000.pdf